CLINICAL TRIAL: NCT07191535
Title: A Multinational Randomized Double-Blind Placebo-Controlled Phase 2 Study to Evaluate the Effect of Linvemastat (FP-020) in Patients With Partially Controlled Asthma on Inhaled Corticosteroids and Long-Acting Beta-Agonists (syMMPonia Study)
Brief Title: Effect of Linvemastat in Patients With Partially Controlled Asthma (syMMPonia)
Acronym: syMMPonia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Collaborators: QPS Holdings LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FP-020C-25-001
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Asthma (Diagnosis); Pulmonary Function; Moderate-to-Severe Asthma
Keywords: central spirometry; type-2 (T2) high asthma; asthma management
MeSH Terms: conditions — Asthma; Disease

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study drug will be provided in bottles. Each bottle contains 32 capsules as a 28-day study drug supply. A bottle is intended for one month (28 days) use with 4 extra capsules allowing for the visit windows and flexibility. Each bottle will have a unique number which is assigned to the study patient by the Interactive Response Technology (IRT) system. All study drugs will be dispensed by the Investigator or a person under his/her supervision
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- linvemastat 100 mg once daily (Experimental): linvemastat 100 mg once daily
  Interventions: Drug: linvemastat
- linvemastat 300 mg once daily (Experimental): linvemastat 300 mg once daily
  Interventions: Drug: linvemastat
- Placebo Comparator (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: linvemastat — Matrix Metalloproteinase-12 inhibitor
  Other Names: FP-020
  Arms: linvemastat 100 mg once daily; linvemastat 300 mg once daily
Drug: Placebo — Placebo
  Arms: Placebo Comparator

SUMMARY:
This study explores a potential new treatment for adults with moderate-to-severe asthma using a drug called linvemastat, which targets an enzyme linked to lung inflammation. Despite using standard asthma medications, many patients still struggle with symptoms, so researchers are testing whether linvemastat can improve lung function and reduce flare-ups. In a carefully controlled trial, participants receive either one of two doses of the drug or a placebo, while continuing their usual treatments. Over 16 weeks, scientists monitor breathing capacity, symptom control, and safety to determine if linvemastat could offer a meaningful new option for asthma management.

DETAILED DESCRIPTION:
This clinical study investigates the potential of a new drug, linvemastat, to improve outcomes for adults with moderate-to-severe asthma who continue to experience symptoms despite using standard treatments like inhaled corticosteroids and long-acting beta-agonists. Linvemastat works by blocking an enzyme called MMP-12, which is believed to contribute to lung inflammation and tissue damage in asthma. The trial is a Phase 2, randomized, double-blind, placebo-controlled study involving approximately 135 participants across multiple global sites. Participants are assigned to receive either 100 mg or 300 mg of linvemastat, or a placebo, once daily for 16 weeks, while continuing their regular asthma medications. Researchers are primarily measuring changes in lung function, specifically the amount of air a person can forcefully exhale in one second (FEV₁), as well as tracking asthma flare-ups, use of rescue inhalers, and markers of inflammation. Safety is closely monitored through lab tests, heart monitoring, and physical exams. The goal is to determine whether linvemastat can offer a meaningful new option for patients whose asthma remains difficult to control, potentially improving both respiratory health and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 85 years at the time of signing informed consent
* Patient is able to provide written informed consent.
* Documented physician´s diagnosis of Type 2 high asthma, as per the Global Initiative for Asthma (GINA) 2023 guideline 2023 at Screening.
* Patients with existing treatment with at least low to medium doses of ICS therapy in combination with LABA as a second controller for at least 90 days and a stable/optimized dose ≥30 days prior to Day 1. Patients on triple therapy with a long-acting muscarinic antagonist (LAMA) will be excluded.
* An ACQ score ≥ 1.5 at Screening.
* Patients with a pre-bronchodilator FEV1 value of 40% to 80% of the patient's predicted value at Screening.
* Patients must have experienced at least once, within 2 years prior to Screening, one of the following asthma exacerbation events: Treatment with a systemic steroid (oral or parenteral) for worsening asthma. Hospitalization or emergency medical care visit for worsening asthma.
* Males with a partner of childbearing potential must use a condom for the duration of study treatment and at least 96 hours after discontinuing the study drug.
* Female patients of childbearing potential (including those < 1 year post-menopausal) must use a highly effective method of contraception per Clinical Trial Facilitation Group (CTFG) recommendation during the conduct of the study and for 30 days after the last dose of study drug. Highly effective contraceptive measures for female patients of childbearing potential include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal. Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable. intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (when partner is the sole sexual partner of the female patient and when the partner has received medical assessment of the surgical success), sexual abstinence.
* Women not of childbearing potential are defined as: Post-menopausal women (defined as at least 12 months with no menses without an alternative medical cause); in women <45 years of age, a high follicle-stimulating hormone (FSH) level in the post-menopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy; OR Have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion at least 6 weeks prior to Screening OR Have a congenital or acquired condition that prevents childbearing.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Current smoker (including vaping) or cessation of smoking within the 6 months prior to Day 1, or > 10 pack-year history of smoking.
* Participation in another clinical trial of an investigational agent within 3 months (small molecule) / 6 months (biologics) or 5 half-lives (if known) of the agent, whichever is longer, prior to randomization.
* Evidence of COVID-19 infection at Screening, as judged by the Investigator.
* Advanced congestive heart failure [New York Heart Association (NYHA) class 3 or 4].
* Known hypersensitivity to any component of the formulation of linvemastat or any component of the excipient.
* Live or messenger ribonucleic acid (mRNA) vaccination within 2 weeks before Day 1 or inoculation with a live or mRNA vaccine is planned during study participation.
* History of solid organ transplant.
* Anti-immunoglobulin E (IgE) therapy [e.g., omalizumab (Xolair®)] within 130 days prior to Screening or any other biologic therapy [including anti-TSLP, anti-IL-4/4R or IL-5/5R monoclonal antibodies (mAb)] or systemic immunosuppressant (e.g., methotrexate) to treat inflammatory disease or autoimmune disease (e.g., rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis) and other diseases, within 2 months or 5 half-lives prior to Screening, whichever is longer.
* Evidence of active tuberculosis (TB) infection at Screening, as judged by the Investigator.
* Active acute or chronic psychiatric illness that, in the opinion of the Investigator, may prevent from complying with study instructions.
* Known positive history of malignancy within 5 years of Screening (with the exception of basal cell skin cancer, carcinoma in-situ of the cervix, or low-risk prostate cancer after curative therapy).
* Positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) infection at Screening.
* Concurrent emphysema.
* Use of any therapeutics that are strong inhibitors and inducers of CYP3A4 or CYP2C8 [e.g., rifampicin, ketoconazole, phenytoin, ritonavir, macrolide antibiotics (e.g., telithromycin), and carbamazepine].
* History of liver dysfunction, including patients with moderate (Child-Pugh B) or severe (Child-Pugh C) impairment or disordered coagulation.
* Abnormal ECG: ventricular arrhythmias (non-sustained ventricular tachycardia [VT], multifocal or frequent premature ventricular contractions, clinically significant bundle branch block or axis deviation [as assessed by PI], or abnormal Q waves). In the case of a corrected QT interval using Fridericia's formula (QTcF) interval >450 ms (men) or >480 ms (women; patients with bundle branch block) or PR (P to QRS) interval outside the range of 120 to 220 ms, the assessment may be repeated once for eligibility determination at Screening or Baseline.
* Known uncontrolled hypertension or diabetes at the discretion of the Investigator.
* Any condition that required hospitalization (except for asthma exacerbation) within the 3 months prior to Day 1 or is likely to require so during the study.
* Clinically significant abnormalities in the Screening physical examination, medical history, vital signs, ECG, or clinical laboratory tests that are not known to be due to concurrent asthma in the opinion of the Investigator and Medical Monitor should preclude the patient's participation in the clinical study.
* The following laboratory parameters are excluded:

  1. Hemoglobin (Hg) <10 g/dL (100 g/L)
  2. White blood cells (WBC) < 3000/μL (< 3000/mm3). African American patients who are known to have low WBC of < 3000/μL but ≥ 1500/μL will be eligible.
  3. Platelet count < 70,000/μL (70,000/mm3)
  4. Serum creatinine > 1.5 x upper limit of normal (ULN)
  5. Glomerular filtration rate ≤ 60 mL/min/1.73 m2 or evidence of acute kidney injury or history of severe hypersensitivity reactions to gadolinium-based contrast agents
  6. Serum total bilirubin > 1.5 ULN
  7. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x ULN or serum alkaline phosphatase > 2 x ULN

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
The mean change in trough FEV1 assessed by central spirometry | Baseline to Week 16
  FEV1 (measured in liters by spirometer), and the trough measurement is taken 24 hours after the morning dose on the previous day of the randomized study drug.
  The Baseline is defined as the last available FEV1 measurement taken prior to the first dose of the randomized study drug.

SECONDARY OUTCOMES:
Time to first severe asthma exacerbation | Baseline up to Week 16].
  Time to first severe asthma exacerbation
Change in clinical laboratory testing | Baseline to Week 16
  Change in mean blood eosinophil count.
FeNO Changes | Baseline up to Week 16
  Change in mean Fraction Exhaled Nitric Oxide (FeNO).
Change in Sputum | Baseline up to Week 16
  Change in mean percentage of mucous eosinophils and neutrophils assessed by sputum analysis
Pre-bronchodilator FEV1 changes | Baseline to Week 16
  Change in mean pre-bronchodilator FEV1.
Post-bronchodilator FEV1 changes | Baseline up to Week 16
  Change in mean post-bronchodilator FEV1.
AM/PM Peak Flow changes | Baseline up to Week 16
  Change in the mean morning and evening Peak Flow (in liters/minute).
Use of Inhaled Corticosteroids (ICS) or Long-Acting Beta-Agonists (LABA) | Baseline to Week 16
  Change in the mean number of inhalations/days of ICS or LABA.
Change in Asthma Control Questionnaire | Baseline up to Week 16
  Change in ACQ score
Change in St. George's Respiratory Questionnaire | Baseline to Week 16
  Change in St. George's Respiratory Questionnaire (SGRQ) score.
Change in clinical laboratory testing | Baseline to Week 16
  Change in mean neutrophil count
Change in clinical laboratory testing | Baseline to Week 16
  Change in mean level of IgE.

CONTACTS AND LOCATIONS:
Overall Officials: Bassem Elmankabadi, MD, Study Director — Foresee Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No